CLINICAL TRIAL: NCT06814561
Title: Hemodynamic Determinants of Urine Output During Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu (Other)
Responsible Party: Principal Investigator, Balan Ion Cosmin, Principal Investigator, Institutul de Urgenţă pentru Boli Cardiovasculare Prof.Dr. C.C. Iliescu
Other Study IDs: 2511
Record Dates: First submitted 2025-02-01; First posted 2025-02-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Urine Output Decreased
Keywords: urine output; spinal anesthesia; mean arterial pressure
MeSH Terms: conditions — Oliguria | interventions — Bupivacaine; Solutions; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Marcaine 0.5% Solution for Injection — The study involves the administration of 0.5% Marcaine heavy for spinal anesthesia in patients undergoing vascular surgery. The aim is to assess how this anesthesia affects urine output relative to mean arterial pressure.
  Other Names: Bupivacaine

SUMMARY:
This clinical trial investigates the relationship between urine output and mean arterial pressure (MAP) during spinal anesthesia. The study aims to validate observations from animal models in humans by concurrently measuring hemoglobin levels, MAP, and urine output, focusing on the effects of Ringer's solution, to provide crucial insights into optimal fluid management during anesthesia with minimal complexity.

DETAILED DESCRIPTION:
The proposed clinical trial aims to explore the relationship between urine output and mean arterial pressure (MAP) during spinal anesthesia, a subject that has not been thoroughly studied in humans despite previous research under general anesthesia. Studies have demonstrated that the diuretic response to intravenous volume loading, using Ringer's solution or 20% albumin, varies with MAP levels. Specifically, Ringer's solution shows a greater diuretic effect when MAP exceeds 70 mmHg, whereas 20% albumin is more effective at lower pressures. This differential response highlights the importance of considering MAP in the choice of fluid for managing hypovolemia and oliguria.

The study's relevance is highlighted by the physiological dynamics at play, particularly how high levels of anesthesia, which influence the sympathetic nervous system from the mid-thoracic region, might reduce MAP and consequently decrease urine output. While this hypothesis has been examined in animal studies, its validity in humans remains unconfirmed.

To address this, the trial will measure hemoglobin levels, MAP, and urine output simultaneously, aiming to establish a clear correlation among these variables during spinal anesthesia. This methodical approach seeks to yield significant insights with minimal additional effort, contrasting with the complexities inherent in more elaborate study designs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by patients or their legally authorized representatives.
* Adults aged 18 years and older.

Exclusion Criteria:

* Contraindications to Spinal Anesthesia:

  * Patient refusal
  * Presence of coagulopathy.
  * Current use of anticoagulant or antiplatelet medications.
  * Critical or severe aortic stenosis or other fixed cardiac output states.
  * High risk of infection at the spinal needle insertion site.
  * Elevated intracranial pressure.
  * Allergy
  * Sepsis
* Procedures Not Amenable to Spinal Anesthesia:

  * Planned concurrent procedures that cannot be performed under spinal anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring spinal anesthesia for vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Catheter-Assisted Urine Output Measurement Post-Spinal Anesthesia | 10, 20, 30, 40, 50, and 60 minutes post-surgical intervention.
  Urine volume is accurately measured using a catheter connected to a graduated collection bag. This method tracks the accumulated volume at specific intervals, providing a precise assessment of renal function and fluid management efficacy following spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hahn, Professor, Study Chair — Karolinska Institutet: Stockholm, SE (Department of Clinical Sciences, Danderyd Hospital) Employment; Serban-Ion Bubenek-Turconi, Professor, Study Director — CC Iliescu Cardiovascular Institute
Locations (1):
- "Prof CC Iliescu" Emergency Institue for Cardiovascular Diseases, Bucharest, Romania